CLINICAL TRIAL: NCT02747992
Title: Comparisons the Analgesia of Paravertebral Block Combined With Thoracic Wall Block Versus Paravertebral Block Alone for Modified Radical Mastectomy in Breast Cancer
Brief Title: Paravertebral Block (PVB) Combined Pectoral Musculature Blocks for Modified Radical Mastectomy (MRM)
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Nai Liang Li, Dr, Sun Yat-sen University
Other Study IDs: PVBPEC
Record Dates: First submitted 2016-04-17; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Mastectomy, Modified Radical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- PECS 0: receiving paravertebral block
- PECS 1: receiving paravertebral block and blocks targeting pectoral musculature

SUMMARY:
Previous studies have shown that PVB reduces pain and postoperative nausea and vomiting after breast cancer surgery when used in addition to general anesthesia or sedation. However, major breast cancer surgery involves areas beyond the breast tissue, such as pectoral musculature.

ELIGIBILITY:
Inclusion Criteria:

* The American Society of Anesthesiologists (ASA) Physical Status classification I to III
* 20 - 75 years of age
* female gender

Exclusion Criteria:

* body mass index (BMI) ≥ 35 kg/m2
* modified radical mastectomy not performed by the single surgeon (Ben Long Yu)
* anesthesia not performed by the single anesthesiologist (Nai Liang Li)

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients were that diagnosed to have unilateral breast cancer and undergone modified radical mastectomy using regional anesthesia during Jun 1, 2012 and May 31, 2015.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
intraoperative sedation requirement | during operation
  target controlled infusion (TCI) propofol driven by the Schnider model in effect site control titrated to reach conscious sedation defined as Observer Assessment of Alertness/Sedation score of 2 to 3

SECONDARY OUTCOMES:
time to first request of analgesics | postoperative 12 hours
postoperative analgesic requirement | postoperation to discharge
side effects | postoperation to within 24 hours after discharge